CLINICAL TRIAL: NCT03308942
Title: Phase 2, Multi-Arm Study of Niraparib Administered Alone and in Combination With a PD-1 Inhibitor in Patients With Non-Small Cell Lung Cancer
Brief Title: Effects of Single Agent Niraparib and Niraparib Plus Programmed Cell Death-1 (PD-1) Inhibitors in Non-Small Cell Lung Cancer Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 213352; 3000-02-001 (Other: Tesaro)
Record Dates: First submitted 2017-10-03; First posted 2017-10-13 (Actual); Results first posted 2021-07-07 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Neoplasms
Keywords: Niraparib; NSCLC; Pembrolizumab; Dostarlimab; TSR-042
MeSH Terms: conditions — Neoplasms | interventions — niraparib; pembrolizumab; dostarlimab

STUDY DESIGN:
Intervention Model Description: Participants will receive niraparib either as monotherapy or in combination with pembrolizumab during Stage 1 of the study. Participants will receive niraparib in combination with TSR-042 (dostarlimab) during Stage 2 of the study.
Masking Description: This will be an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Stage 1 (Cohort 1): Niraparib plus Pembrolizumab (Experimental): Participants with locally advanced and metastatic NSCLC (all histologies) with no prior systemic chemotherapy or PD-1/programmed death-ligand 1 (PD-L1) inhibitor treatment and whose tumors have high PD-L1 expression (tumor proportion score [TPS]: >= 50 percent [%]) will receive combination of niraparib and a PD-1 inhibitor; pembrolizumab.
  Interventions: Drug: Niraparib; Biological: Pembrolizumab
- Stage 1 (Cohort 2): Niraparib plus Pembrolizumab (Experimental): Participants with locally advanced and metastatic NSCLC (all histologies) with no prior systemic chemotherapy or PD-1/PD-L1 inhibitor treatment and whose tumors have PD-L1 expression (TPS: 1% to 49%) will receive combination of niraparib and a PD-1 inhibitor; pembrolizumab.
  Interventions: Drug: Niraparib; Biological: Pembrolizumab
- Stage 1 (Cohort 3): Niraparib (Experimental): Participants with locally advanced and metastatic squamous NSCLC who have been previously treated with both platinum and either PD-1 or PD-L1 inhibitor will receive single agent niraparib.
  Interventions: Drug: Niraparib
- Stage 2 (Cohort 1A): Niraparib plus TSR-042 (Dostarlimab) (Experimental): Participants with locally advanced and metastatic NSCLC (all histologies) with no prior systemic chemotherapy or PD-1/PD-L1 inhibitor treatment and whose tumors have high PD-L1 expression (TPS: >= 50%) will receive combination of niraparib and a PD-1 inhibitor; TSR-042 (Dostarlimab).
  Interventions: Drug: Niraparib; Biological: TSR-042 (Dostarlimab)
- Stage 2 (Cohort 2A): Niraparib plus TSR-042 (Dostarlimab) (Experimental): Participants with locally advanced and metastatic NSCLC (all histologies) with no prior systemic chemotherapy or PD-1/PD-L1 inhibitor treatment and whose tumors have PD-L1 expression (TPS: 1% to 49%) will receive combination of niraparib and a PD-1 inhibitor; TSR-042 (Dostarlimab).
  Interventions: Drug: Niraparib; Biological: TSR-042 (Dostarlimab)

INTERVENTIONS:
Drug: Niraparib — Niraparib is an orally available, potent, highly selective poly adenosine diphosphate- ribose (poly ADP-ribose) polymerase-1 (PARP-1) and PARP-2 inhibitor. It will be available as 100 milligrams (mg) capsules and will be administered as 2 X 100 mg capsules (200 mg per day) orally once daily (QD).
Biological: Pembrolizumab — Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the immunoglobulin G-4 (IgG4)/kappa isotype designed to directly block the interaction between PD-1 and its ligands (PD-L1 and PD-L2). It will be available as 50 mg lyophilized powder single-use vials or 100 mg/4 milliliters (mL) (25 mg/mL) solution in a single-dose vial. It will be administered at a dose of 200 mg intravenous (IV) using a 30-minute IV infusion
  Arms: Stage 1 (Cohort 1): Niraparib plus Pembrolizumab; Stage 1 (Cohort 2): Niraparib plus Pembrolizumab
Biological: TSR-042 (Dostarlimab) — TSR-042 (Dostarlimab) is a humanized mAb of the IgG4/kappa isotype that binds with high affinity to PD-1, resulting in inhibition of binding to PD-L1 and PD-L2. It will be administered at a dose of 500 mg for every 3 weeks (Q3W) for first 4 cycles followed by 1000 mg for every 6 weeks (Q6W) for all subsequent cycles using a 30-minute IV infusion. TSR-042 (dostarlimab) will be supplied as a solution of 160 mg (20 mg/mL) or 500 mg (50 mg/mL) in a single-dose vial.
  Arms: Stage 2 (Cohort 1A): Niraparib plus TSR-042 (Dostarlimab); Stage 2 (Cohort 2A): Niraparib plus TSR-042 (Dostarlimab)

SUMMARY:
This is a multicenter, open-label, phase 2 study to evaluate the efficacy and safety of niraparib alone and in combination with PD-1 inhibitors in participants with locally advanced and metastatic non-small cell lung cancer (NSCLC). The study will consist of 2 stages. In stage 1, participants from Cohorts 1 and 2 will receive niraparib plus PD-1 inhibitor; pembrolizumab and participants from Cohort 3 will receive niraparib alone. In Stage 2, participants from Cohorts 1A and 2A will receive niraparib plus the PD-1 inhibitor, TSR-042 (Dostarlimab).

ELIGIBILITY:
General Inclusion Criteria:

* Male or female participants at least 18 years of age.
* Histological or cytological proven advanced (unresectable) or metastatic NSCLC as defined as stage IIIB (positive supraclavicular lymph nodes) not amenable to definitive chemoradiotherapy or stage IV NSCLC.
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Adequate organ function, defined as:

  1. Absolute neutrophil count (ANC) >= 1500 per microliter (/µL).
  2. Platelets >= 100,000/µL.
  3. Hemoglobin >= 9 grams per deciliter (g/dL) or >= 5.6 millimoles per liter (mmol/L).
  4. Serum creatinine <= 1.5 times upper limit of normal (ULN) or creatinine clearance >= 50 milliliters per minute (mL/min) (as calculated using the Cockcroft Gault equation or measured using 24-hour urine creatinine clearance) for participants with creatinine levels > 1.5 times institutional ULN.
  5. Total bilirubin <= 1.5 times ULN except in participants with Gilbert's syndrome. Participants with Gilbert's syndrome may enroll if direct bilirubin <= 1.5 times ULN of the direct bilirubin.
  6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 2.5 times ULN unless liver metastases are present, in which case they must be <= 5 times ULN.
* Participant must have recovered to Grade 1 toxicity from prior cancer therapy (a participant with Grade 2 neuropathy or Grade 2 alopecia is an exception to this criterion and may qualify for this study).
* Participant agrees to submit formalin fixed paraffin embedded (FFPE) tumor tissue specimen, which may have been collected at any time prior to screening. If no archival FFPE tumor tissue is available, participant agrees to undergo a tumor tissue biopsy before Cycle 1/Day 1. (For Cohort 3 only: if diagnosis was made by cytology and archival tissue is not available, participant will not need to provide tumor tissue).
* Participants is able to take oral medications.
* Female participant meets the following criteria:

  a) Female participant (of childbearing potential) is not breastfeeding, has a negative serum pregnancy test within 72 hours prior to taking study drug, and agrees to abstain from activities that could result in pregnancy from enrollment through 180 days after the last dose of study treatment or is of nonchildbearing potential; or b) Female participant is of nonchildbearing potential, other than medical reasons, defined as follows: i) >=45 years of age and has not had menses for > 1 year. ii) Amenorrheic for < 2 years without a hysterectomy and oophorectomy and a follicle-stimulating hormone (FSH) value in the postmenopausal range upon screening evaluation.

iii) Post hysterectomy, bilateral oophorectomy, or tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the participant must be willing to use 2 highly effective contraception methods throughout the study, starting with the screening visit through 180 days after the last dose of study therapy.

* Male participant agrees to use an adequate method of contraception and not donate sperm starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Participant is able to understand the study procedures and agree to participate in the study by providing written informed consent.

Cohort Specific Inclusion Criteria:

* Cohorts 1 and 1A (combination of niraparib and PD-1 inhibitor): participants must have tumors with high PD-L1 expression (TPS >= 50%) per local assessment; with no known Epidermal Growth Factor Receptor (EGFR)-sensitizing mutation and/or ROS -1 or anaplastic lymphoma kinase (ALK) translocation, and no prior systemic chemotherapy or PD-1/PD-L1 inhibitor treatment for metastatic NSCLC.
* Cohorts 2 and 2A (combination of niraparib and PD-1 inhibitor): participants must have tumors with PD-L1 expression (TPS between 1% and 49%) per local assessment, with no known EGFR-sensitizing mutation and/or ROS-1 or ALK translocation, and no prior systemic chemotherapy or PD-1/PD-L1 inhibitor treatment for metastatic NSCLC.
* Cohort 3 (single agent niraparib): participants must have metastatic squamous non-small cell lung cancer (sqNSCLC) and have progressed after both prior platinum-based chemotherapy and prior PD-1 or PD-L1 inhibitor treatment.

Exclusion Criteria for Cohorts 1, 1A , 2 and 2A:

* Participant has received systemic therapy for the treatment of advanced stage NSCLC. Completion of treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of metastatic disease.
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Known hypersensitivity to the components of niraparib, pembrolizumab, TSR-042 (Dostarlimab), or their excipients.
* Known EGFR (exon 19 and 21) mutations, ALK translocations, and/or ROS-1 translocations.
* Participant has a history or current condition (such as transfusion-dependent anemia or thrombocytopenia), therapy, or laboratory abnormality that might confound the study results, or interfere with the participant's participation for the full duration of the study treatment.
* Known diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
* Participant is immunocompromised, in the opinion of the Investigator.
* Current participation in a treatment study or past participation in a study of an investigational agent within 4 weeks before the first dose of study treatment.
* Symptomatic uncontrolled brain or leptomeningeal metastases. (To be considered "controlled," central nervous system [CNS] disease must have undergone treatment [example, radiation or chemotherapy] at least 1 month prior to study entry. The participant must not have any new or progressive signs or symptoms related to the CNS disease and must be taking <= 10 mg of prednisone or equivalent per day or no steroids.) Participants who have untreated brain metastases and who are not symptomatic may enroll if the Investigator feels that treatment of these metastases is not indicated. A scan to confirm the absence of brain metastases is not required. Participants with spinal cord compression may be considered if they have received definitive treatment for this and evidence of clinically SD for 28 days.
* Active autoimmune disease that required systemic treatment in the past 2 years (with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (examples, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Major surgery within 3 weeks of starting the study or participant has not recovered from any effects of any major surgery.
* Other active concomitant malignancy that warrants systemic therapy.
* Poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, uncontrolled hypertension, active uncontrolled coagulopathy or any psychiatric disorder that prohibits obtaining informed consent.
* Known history of interstitial lung disease, drug-related pneumonitis, or radiation pneumonitis requiring steroid treatment.
* Participant is pregnant, breastfeeding, or expecting to conceive children while receiving study treatment and for 180 days (for pregnancy or conception) or 30 days (for breastfeeding) after the last dose of study treatment.
* Male participant is expecting to donate sperm or father children while receiving study drug or for 120 days after the last dose of study treatment.
* Known active hepatic disease (known hepatic cirrhosis, hepatitis B surface antigen-positive status, or suspected active hepatitis C infection).
* Prior treatment with a known poly adenosine diphosphate-ribose (ADP-ribose) polymerase (PARP) inhibitor.
* Participant received a live vaccine within 30 days of planned start of study therapy.
* Known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).

Exclusion criteria for Cohort 3:

* Platinum-treated participant who progressed while on or within less than 8 weeks from the last day of platinum administration.
* Known hypersensitivity to the components of niraparib or excipients.
* Participant has a history or current condition (such as transfusion dependent anemia or thrombocytopenia), therapy, or laboratory abnormality that might confound the study results, or interfere with the participant's participation for the full duration of the study treatment.
* Known diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
* Current participation in a treatment study or past participation in a study of an investigational agent within 4 weeks before the first dose of study treatment.
* Symptomatic uncontrolled brain or leptomeningeal metastases. (To be considered "controlled," CNS disease must have undergone treatment [example, radiation or chemotherapy] at least 1 month prior to study entry. The participant must not have any new or progressive signs or symptoms related to the CNS disease and must be taking <= 10 mg of prednisone or equivalent per day or no steroids.) Participants who have untreated brain metastases and who are not symptomatic may enroll if the investigator feels that treatment of these metastases is not indicated. A scan to confirm the absence of brain metastases is not required. Participants with spinal cord compression may be considered if they have received definitive treatment for this and evidence of clinically SD for 28 days.
* Major surgery within 3 weeks of starting the study or participant has not recovered from any effects of any major surgery.
* Other active concomitant malignancy that warrants systemic therapy.
* Poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, uncontrolled hypertension, active uncontrolled coagulopathy, or any psychiatric disorder that prohibits obtaining informed consent.
* Known history of interstitial lung disease, drug-related pneumonitis, or radiation pneumonitis requiring steroid treatment.
* Participant is pregnant, breastfeeding, or expecting to conceive children, while receiving study treatment and for 180 days (for pregnancy or conception) or 30 days (for breastfeeding) after the last dose of study treatment.
* Male participant is expecting to donate sperm or father children while receiving study drug or for 120 days after the last dose of study treatment.
* Participant is immunocompromised, in the opinion of the Investigator.
* Known active hepatic disease (known hepatic cirrhosis, hepatitis B surface antigen-positive status, or suspected active hepatitis C infection).
* Prior treatment with a known PARP inhibitor.
* Known history of MDS or AML.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- United States (16):
  - GSK Investigational Site, Whittier, Alaska
  - GSK Investigational Site, Port Saint Lucie, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Harvey, Illinois
  - GSK Investigational Site, Tinley Park, Illinois
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Florham Park, New Jersey
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Kennewick, Washington
  - GSK Investigational Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency

REFERENCES:
- [Background] Ramalingam SS, Thara E, Awad MM, Dowlati A, Haque B, Stinchcombe TE, Dy GK, Spigel DR, Lu S, Iyer Singh N, Tang Y, Teslenko I, Iannotti N. JASPER: Phase 2 trial of first-line niraparib plus pembrolizumab in patients with advanced non-small cell lung cancer. Cancer. 2022 Jan 1;128(1):65-74. doi: 10.1002/cncr.33885. Epub 2021 Sep 3. PMID 34478166

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of two stages; Stage 1 (Cohorts 1, 2, 3) and Stage 2 (Cohorts 1A, 2A).
Pre-assignment Details: A total of 69 participants were screened, of which 16 failed screening and 53 participants (41 in Stage 1 and 12 in Stage 2) were enrolled into the study. Data was not collected for Cohort 2A of Stage 2 as the Sponsor decided not to open this Cohort to enrollment.
Groups:
- Stage 1 (Cohort 1): Niraparib + Pembrolizumab: Participants with locally advanced and metastatic non-small cell lung cancer (NSCLC) (all histologies) with no prior systemic chemotherapy or programmed cell death-1 (PD-1)/programmed death-ligand 1 (PD-L1) inhibitor treatment and whose tumors had high PD-L1 expression (tumor proportion score [TPS]: >= 50 percent [%]) received a combination of niraparib and pembrolizumab. Niraparib was given at a dose of 200 milligrams (mg) orally once daily during each 21-day cycle. Pembrolizumab was administered as an intravenous (IV) infusion at a dose of 200 mg on Day 1 of each 21-day cycle.
- Stage 1 (Cohort 2): Niraparib + Pembrolizumab: Participants with locally advanced and metastatic NSCLC (all histologies) with no prior systemic chemotherapy or PD-1/PD-L1 inhibitor treatment and whose tumors had PD-L1 expression (TPS: 1% to 49%) received a combination of niraparib and pembrolizumab. Niraparib was given at a dose of 200 mg orally once daily during each 21-day cycle. Pembrolizumab was administered as an IV infusion at a dose of 200 on Day 1 of each 21-day cycle.
- Stage 1 (Cohort 3): Niraparib: Participants with locally advanced and metastatic squamous NSCLC who were previously treated with both platinum and either PD-1 or PD-L1 inhibitor received single agent niraparib at a dose of 200 mg orally once daily during each 21-day cycle.
- Stage 2 (Cohort 1A): Niraparib + TSR-042 (Dostarlimab): Participants with locally advanced and metastatic NSCLC (all histologies) with no prior systemic chemotherapy or PD-1/PD-L1 inhibitor treatment and whose tumors have high PD-L1 expression (TPS: >= 50%) received a combination of niraparib and TSR-042 (Dostarlimab). Niraparib was given at a dose of 200 mg orally once daily during each 21-day cycle. TSR-042 (Dostarlimab) was administered as an IV infusion at a dose of 500 mg once every 3 weeks for first 4 cycles followed by 1000 mg dose once every 6 weeks for subsequent cycles (each cycle of 21 days).
- Stage 2 (Cohort 2A): Niraparib + TSR-042 (Dostarlimab): Participants with locally advanced and metastatic NSCLC (all histologies) with no prior systemic chemotherapy or PD-1/PD-L1 inhibitor treatment and whose tumors have PD-L1 expression (TPS: 1% to 49%) were planned to receive a combination of niraparib and TSR-042 (Dostarlimab). Niraparib was planned to be given at a dose of 200 mg orally once daily. TSR-042 (Dostarlimab) was planned to be administered as an IV infusion at a dose of 500 mg once every 3 weeks for first 4 cycles followed by 1000 mg dose once every 6 weeks for all subsequent cycles (each cycle of 21 days).
Period: Stage 1 (Up to a Maximum of 45 Months)
Arm/Group | Stage 1 (Cohort 1): Niraparib + Pembrolizumab | Stage 1 (Cohort 2): Niraparib + Pembrolizumab | Stage 1 (Cohort 3): Niraparib | Stage 2 (Cohort 1A): Niraparib + TSR-042 (Dostarlimab) | Stage 2 (Cohort 2A): Niraparib + TSR-042 (Dostarlimab)
Started | 17 | 21 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 17 | 21 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 2 | 0 | 0
Not completed — Death | 11 | 16 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Sponsor Decision | 3 | 1 | 0 | 0 | 0
Period: Stage 2 (Up to a Maximum of 29 Months)
Arm/Group | Stage 1 (Cohort 1): Niraparib + Pembrolizumab | Stage 1 (Cohort 2): Niraparib + Pembrolizumab | Stage 1 (Cohort 3): Niraparib | Stage 2 (Cohort 1A): Niraparib + TSR-042 (Dostarlimab) | Stage 2 (Cohort 2A): Niraparib + TSR-042 (Dostarlimab)
Started | 0 | 0 | 0 | 12 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 12 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 0
Not completed — Death | 0 | 0 | 0 | 6 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Data was not collected for Cohort 2A of Stage 2 as no participant was enrolled into this Cohort of the study. Safety Population comprised of participants who received at least one dose of either study medications.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1 (Cohort 1): Niraparib + Pembrolizumab | Stage 1 (Cohort 2): Niraparib + Pembrolizumab | Stage 1 (Cohort 3): Niraparib | Stage 2 (Cohort 1A): Niraparib + TSR-042 (Dostarlimab) | Stage 2 (Cohort 2A): Niraparib + TSR-042 (Dostarlimab) | Total
Number analyzed (Participants) | 17 | 21 | 3 | 12 | 0 | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.1 (7.55) | 70.9 (9.78) | 72.3 (10.69) | 68.3 (6.74) |  | 70.1 (8.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 0 | 6 |  | 24
  Male | 11 | 9 | 3 | 6 |  | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 |  | 1
  Asian | 0 | 1 | 0 | 1 |  | 2
  Black or African American | 1 | 0 | 0 | 2 |  | 3
  White | 14 | 19 | 3 | 8 |  | 44
  Unknown | 2 | 1 | 0 | 0 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Cohort 1: Objective Response Rate (ORR)
Description: ORR is the percentage of participants with a confirmed best overall response (BOR) of complete response (CR) or partial response (PR) in the analysis population where CR=Disappearance of all target lesions. Any pathological lymph nodes must be <10 millimeters (mm) in the short axis. PR=At least a 30 percent (%) decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters. Tumor assessment was done by the Investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. Data has been presented for participants with NSCLC whose tumors have high PD-L1 expression (TPS>=50%). Confidence interval was calculated using binomial exact method.
Time Frame: Up to a maximum of 29 months
Population: Modified intent-to-treat (mITT) Population comprised of all participants who received any study drug and did not withdraw consent prior to having at least one post-Baseline tumor assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 1 (Cohort 1): Niraparib + Pembrolizumab
Number analyzed (Participants) | 16
Percentage of participants | 56.3 [29.9 to 80.2]

2. Primary Outcome: Stage 1: Cohort 2: Objective Response Rate
Description: ORR is the percentage of participants with a confirmed BOR of CR or PR in the analysis population where CR=Disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis. PR=At least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters. Tumor assessment was done by the Investigator per RECIST v1.1. Data has been presented for participants with NSCLC having PD-L1 expression in tumors (TPS: 1 to 49%). Confidence interval was calculated using binomial exact method.
Time Frame: Up to a maximum of 17 months
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 1 (Cohort 2): Niraparib + Pembrolizumab
Number analyzed (Participants) | 20
Percentage of participants | 20.0 [5.7 to 43.7]

3. Primary Outcome: Stage 1: Cohort 3: Objective Response Rate
Description: ORR is the percentage of participants with a confirmed BOR of CR or PR in the analysis population where CR=Disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis. PR=At least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters. Tumor assessment was done by the Investigator per RECIST v1.1. Data is presented for participants with locally advanced and metastatic squamous NSCLC. Confidence interval was calculated using binomial exact method.
Time Frame: Up to a maximum of 6 months
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 1 (Cohort 3): Niraparib
Number analyzed (Participants) | 2
Percentage of participants | 0 [0.0 to 84.2]

4. Primary Outcome: Stage 2: Cohort 1A and Cohort 2A: Objective Response Rate
Description: ORR is the percentage of participants with a confirmed BOR of CR or PR in the analysis population where CR=Disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis. PR=At least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters. Tumor assessment was done by the Investigator per RECIST v1.1. Confidence interval was calculated using binomial exact method.
Time Frame: Up to a maximum of 17 months
Population: mITT Population. Data was not collected for Cohort 2A of Stage 2 as no participant was enrolled into this Cohort of the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Stage 2 (Cohort 2A): Niraparib + TSR-042 (Dostarlimab): Participants with locally advanced and metastatic NSCLC (all histologies) with no prior systemic chemotherapy or PD-1/PD-L1 inhibitor treatment and whose tumors have PD-L1 expression (TPS: 1% to 49%) were planned to receive a combination of niraparib and TSR-042 (Dostarlimab). Niraparib was planned to be given at a dose of 200 mg orally once daily. TSR-042 (Dostarlimab) was planed to be administered as an IV infusion at a dose of 500 mg once every 3 weeks for first 4 cycles followed by 1000 mg dose once every 6 weeks for all subsequent cycles (each cycle of 21 days).
Arm/Group | Stage 2 (Cohort 1A): Niraparib + TSR-042 (Dostarlimab) | Stage 2 (Cohort 2A): Niraparib + TSR-042 (Dostarlimab)
Number analyzed (Participants) | 11 | 0
Percentage of participants | 9.1 [0.2 to 41.3] |

5. Secondary Outcome: Stage 1: Cohort 1: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence that occurs in a participant or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with this treatment. A SAE is defined as any untoward medical occurrence that, at any dose that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, is an important medical event(s) as per medical and scientific judgment. Adverse events which were not Serious Adverse Events were considered as Non-Serious adverse events
Time Frame: Up to a maximum of 45 months
Population: Safety Population comprised of participants who received at least one dose of either study medications.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (Cohort 1): Niraparib + Pembrolizumab
Number analyzed (Participants) | 17
Participants
  Any SAE | 11
  Any non-SAE | 17

6. Secondary Outcome: Stage 1: Cohort 2: Number of Participants With Non-SAEs and SAEs
Description: An AE is any untoward medical occurrence that occurs in a participant or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with this treatment. A SAE is defined as any untoward medical occurrence that, at any dose that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, is an important medical event(s) as per medical and scientific judgment. Adverse events which were not Serious Adverse Events were considered as Non-Serious adverse events
Time Frame: Up to a maximum of 17 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (Cohort 2): Niraparib + Pembrolizumab
Number analyzed (Participants) | 21
Participants
  Any SAE | 14
  Any non-SAE | 20

7. Secondary Outcome: Stage 1: Cohort 3: Number of Participants With Non-SAEs and SAEs
Description: as for outcome 6
Time Frame: Up to a maximum of 6 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (Cohort 3): Niraparib
Number analyzed (Participants) | 3
Participants
  Any SAE | 1
  Any non-SAE | 3

8. Secondary Outcome: Stage 2: Cohorts 1A and 2A: Number of Participants With Non-SAEs and SAEs
Description: as for outcome 6
Time Frame: Up to a maximum of 29 months
Population: Safety Population. Data was not collected for Cohort 2A of Stage 2 as no participant was enrolled into this Cohort of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 (Cohort 1A): Niraparib + TSR-042 (Dostarlimab) | Stage 2 (Cohort 2A): Niraparib + TSR-042 (Dostarlimab)
Number analyzed (Participants) | 12 | 0
Participants
  Any SAE | 7 |
  Any non-SAE | 12 |

9. Secondary Outcome: Stage 1: Cohort 1: Number of Participants Discontinuing the Study Due to AEs
Description: An AE is any untoward medical occurrence that occurs in a participant or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with this treatment. Number of participants discontinuing the study due to AEs have been summarized.
Time Frame: Up to a maximum of 45 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (Cohort 1): Niraparib + Pembrolizumab
Number analyzed (Participants) | 17
Participants | 10

10. Secondary Outcome: Stage 1: Cohort 2: Number of Participants Discontinuing the Study Due to AEs
Description: as for outcome 9
Time Frame: Up to a maximum of 17 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (Cohort 2): Niraparib + Pembrolizumab
Number analyzed (Participants) | 21
Participants | 9

11. Secondary Outcome: Stage 1: Cohort 3: Number of Participants Discontinuing the Study Due to AEs
Description: as for outcome 9
Time Frame: Up to a maximum of 6 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (Cohort 3): Niraparib
Number analyzed (Participants) | 3
Participants | 1

12. Secondary Outcome: Stage 2: Cohorts 1A and 2A: Number of Participants Discontinuing the Study Due to AEs
Description: as for outcome 9
Time Frame: Up to maximum 29 months
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 (Cohort 1A): Niraparib + TSR-042 (Dostarlimab) | Stage 2 (Cohort 2A): Niraparib + TSR-042 (Dostarlimab)
Number analyzed (Participants) | 12 | 0
Participants | 2 |

13. Secondary Outcome: Stage 1: Cohort 1: Duration of Response
Description: Duration of Response was defined as the time from first documented CR or PR until the subsequently documented disease progression by RECIST v1.1 or death, whichever occurs earlier; where CR=Disappearance of all target lesions. Any pathological lymph nodes must be <10 millimeter (mm) in the short axis. PR=At least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters.
Time Frame: Up to a maximum of 45 months
Population: mITT Population. Only those participants with confirmed response were analyzed.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Stage 1 (Cohort 1): Niraparib + Pembrolizumab
Number analyzed (Participants) | 9
Months | 22.8 [10.1 to NA] — NA indicates <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived.

14. Secondary Outcome: Stage 1: Cohort 2: Duration of Response
Description: Duration of Response was defined as the time from first documented CR or PR until the subsequently documented disease progression by RECIST v1.1 or death, whichever occurs earlier; where CR=Disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis. PR=At least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters.
Time Frame: Up to a maximum of 17 months
Population: mITT Population. Only those participants with confirmed response were analyzed.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Stage 1 (Cohort 2): Niraparib + Pembrolizumab
Number analyzed (Participants) | 4
Months | 9.4 [5.2 to 13.8]

15. Secondary Outcome: Stage 1 : Cohort 3: Duration of Response
Description: as for outcome 14
Time Frame: Up to a maximum of 6 months
Population: mITT Population. No participant had confirmed response. Hence, data for duration of response was not collected.
Arm/Group | Stage 1 (Cohort 3): Niraparib
Number analyzed (Participants) | 0

16. Secondary Outcome: Stage 2: Cohorts 1A and 2A: Duration of Response
Description: as for outcome 14
Time Frame: Up to a maximum of 29 months
Population: mITT Population. Only those participants with confirmed response were analyzed. Data was not collected for Cohort 2A of Stage 2 as no participant was enrolled into this Cohort of the study.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Stage 2 (Cohort 1A): Niraparib + TSR-042 (Dostarlimab) | Stage 2 (Cohort 2A): Niraparib + TSR-042 (Dostarlimab)
Number analyzed (Participants) | 1 | 0
Months | 21.5 [NA to NA] — NA indicates, as there was a single participant, median value presented is the actual value. Hence, inter quartile range could not be calculated for single participant. |

17. Secondary Outcome: Stage 1 : Cohort 1: Disease Control Rate
Description: Disease Control Rate was defined as the percentage of participants with a best overall response of CR, PR or SD per RECIST v1.1; where CR=Disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis. PR=At least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters. Confidence interval was calculated using binomial exact method.
Time Frame: Up to a maximum of 45 months
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 1 (Cohort 1): Niraparib + Pembrolizumab
Number analyzed (Participants) | 16
Percentage of participants | 87.5 [61.7 to 98.4]

18. Secondary Outcome: Stage 1 : Cohort 2: Disease Control Rate
Description: as for outcome 17
Time Frame: Up to a maximum of 17 months
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 1 (Cohort 2): Niraparib + Pembrolizumab
Number analyzed (Participants) | 20
Percentage of participants | 70.0 [45.7 to 88.1]

19. Secondary Outcome: Stage 1 : Cohort 3: Disease Control Rate
Description: as for outcome 17
Time Frame: Up to a maximum of 6 months
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 1 (Cohort 3): Niraparib
Number analyzed (Participants) | 2
Percentage of participants | 50.0 [1.3 to 98.7]

20. Secondary Outcome: Stage 2: Cohorts 1A and 2A: Disease Control Rate
Description: as for outcome 17
Time Frame: Up to a maximum of 29 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 2 (Cohort 1A): Niraparib + TSR-042 (Dostarlimab) | Stage 2 (Cohort 2A): Niraparib + TSR-042 (Dostarlimab)
Number analyzed (Participants) | 11 | 0
Percentage of participants | 54.5 [23.4 to 83.3] |

21. Secondary Outcome: Stage 1 : Cohort 1: Progression-free Survival
Description: Progression-free survival was defined as the time from the date of first dose to the date of disease progression or death due to any cause, whichever occurs earlier. Progression was defined using RECIST v1.1 as a 20% increase in the sum of the diameter of target lesions or unequivocal progression of existing non-target lesions or the appearance of one or more new lesions.
Time Frame: Up to a maximum of 45 months
Population: mITT Population
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Stage 1 (Cohort 1): Niraparib + Pembrolizumab
Number analyzed (Participants) | 16
Months | 8.4 [3.9 to 36.2]

22. Secondary Outcome: Stage 1 : Cohort 2: Progression-free Survival
Description: as for outcome 21
Time Frame: Up to a maximum of 17 months
Population: mITT Population
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Stage 1 (Cohort 2): Niraparib + Pembrolizumab
Number analyzed (Participants) | 20
Months | 4.2 [2.0 to 6.2]

23. Secondary Outcome: Stage 1 : Cohort 3: Progression-free Survival
Description: as for outcome 21
Time Frame: Up to a maximum of 6 months
Population: mITT Population
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Stage 1 (Cohort 3): Niraparib
Number analyzed (Participants) | 2
Months | 4.0 [1.3 to 6.6]

24. Secondary Outcome: Stage 2: Cohorts 1A and 2A: Progression-free Survival
Description: as for outcome 21
Time Frame: Up to a maximum of 29 months
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Stage 2 (Cohort 1A): Niraparib + TSR-042 (Dostarlimab) | Stage 2 (Cohort 2A): Niraparib + TSR-042 (Dostarlimab)
Number analyzed (Participants) | 11 | 0
Months | 4.4 [2.0 to NA] — NA indicates that <55% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived. |

25. Secondary Outcome: Stage 1: Cohort 1: Plasma Concentration of Niraparib Following Combination Therapy of Niraparib and Pembrolizumab
Description: Blood samples were collected at indicated time points.
Time Frame: Cycle 1 Day 1(Pre-dose and 30 Minutes, 1 Hour, 2 Hours, 4 Hours, 8 Hours, 96 Hours, 168 Hours Post-dose); Cycles 2, 4, 8 (Pre-dose and 4 Hours Post-dose) (each cycle of 21 days)
Population: Pharmacokinetic Population comprised of participants who had at least one of measurable niraparib concentration. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Stage 1 (Cohort 1): Niraparib + Pembrolizumab
Number analyzed (Participants) | 17
Nanograms per milliliter
  Cycle 1 Day 1; Pre-dose | 28.4 (115)
  Cycle 1 Day 1; 30 Minutes Post-dose: number analyzed (Participants) | 1
  Cycle 1 Day 1; 30 Minutes Post-dose | 201 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 1 Day 1; 1 Hour Post-dose: number analyzed (Participants) | 1
  Cycle 1 Day 1; 1 Hour Post-dose | 500 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 1 Day 1; 2 Hours Post-dose: number analyzed (Participants) | 1
  Cycle 1 Day 1; 2 Hours Post-dose | 733 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 1 Day 1; 4 Hours Post-dose | 335 (233)
  Cycle 1 Day 1; 8 Hours Post-dose: number analyzed (Participants) | 1
  Cycle 1 Day 1; 8 Hours Post-dose | 353 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 1 Day 1; 96 Hours Post-dose: number analyzed (Participants) | 1
  Cycle 1 Day 1; 96 Hours Post-dose | 1400 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 1 Day 1; 168 Hours Post-dose: number analyzed (Participants) | 1
  Cycle 1 Day 1; 168 Hours Post-dose | 1440 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 2; Pre-dose: number analyzed (Participants) | 12
  Cycle 2; Pre-dose | 360 (383)
  Cycle 2; 4 Hours Post-dose: number analyzed (Participants) | 13
  Cycle 2; 4 Hours Post-dose | 959 (506)
  Cycle 4; Pre-dose: number analyzed (Participants) | 9
  Cycle 4; Pre-dose | 600 (505)
  Cycle 4; 4 Hours Post-dose: number analyzed (Participants) | 10
  Cycle 4; 4 Hours Post-dose | 794 (597)
  Cycle 8; Pre-dose: number analyzed (Participants) | 9
  Cycle 8; Pre-dose | 460 (543)
  Cycle 8; 4 Hours Post-dose: number analyzed (Participants) | 7
  Cycle 8; 4 Hours Post-dose | 727 (824)

26. Secondary Outcome: Stage 1: Cohort 2: Plasma Concentration of Niraparib Following Combination Therapy of Niraparib and Pembrolizumab
Description: Blood samples were collected at indicated time points.
Time Frame: Cycle 1 Day 1 (Pre-dose and 30 Minutes, 1, 2, 4, 8, 24, 168, 336 Hours Post-dose), Cycles 2, 8 (Pre-dose and 4 Hours Post-dose), Cycle 4 (Pre-dose and 30 Minutes, 1, 2, 4, 8, 24, 96, 168, 336 Hours Post-dose) (each cycle of 21 days)
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Stage 1 (Cohort 2): Niraparib + Pembrolizumab
Number analyzed (Participants) | 21
Nanograms per milliliter
  Cycle 1 Day 1; Pre-dose: number analyzed (Participants) | 19
  Cycle 1 Day 1; Pre-dose | NA (NA) — NA indicates that data was not available as no concentration values were detected for pre-dose.
  Cycle 1 Day 1; 30 Minutes Post-dose: number analyzed (Participants) | 3
  Cycle 1 Day 1; 30 Minutes Post-dose | 24.5 (42.4)
  Cycle 1 Day 1; 1 Hour Post-dose: number analyzed (Participants) | 3
  Cycle 1 Day 1; 1 Hour Post-dose | 189 (302)
  Cycle 1 Day 1; 2 Hours Post-dose: number analyzed (Participants) | 3
  Cycle 1 Day 1; 2 Hours Post-dose | 264 (251)
  Cycle 1 Day 1; 4 Hours Post-dose | 345 (188)
  Cycle 1 Day 1; 8 Hours Post-dose: number analyzed (Participants) | 2
  Cycle 1 Day 1; 8 Hours Post-dose | 238 (NA) — NA indicates that standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.
  Cycle 1 Day 1; 24 Hours Post-dose: number analyzed (Participants) | 2
  Cycle 1 Day 1; 24 Hours Post-dose | 318 (NA) — NA indicates that standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.
  Cycle 1 Day 1; 168 Hours Post-dose: number analyzed (Participants) | 1
  Cycle 1 Day 1; 168 Hours Post-dose | 759 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 1 Day 1; 336 Hours Post-dose: number analyzed (Participants) | 1
  Cycle 1 Day 1; 336 Hours Post-dose | 808 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 2; Pre-dose: number analyzed (Participants) | 12
  Cycle 2; Pre-dose | 767 (362)
  Cycle 2; 4 Hours Post-dose: number analyzed (Participants) | 11
  Cycle 2; 4 Hours Post-dose | 1170 (473)
  Cycle 4; Pre-dose: number analyzed (Participants) | 9
  Cycle 4; Pre-dose | 805 (588)
  Cycle 4; 30 Minutes Post-dose: number analyzed (Participants) | 1
  Cycle 4; 30 Minutes Post-dose | 841 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 4; 1 Hour Post-dose: number analyzed (Participants) | 1
  Cycle 4; 1 Hour Post-dose | 1260 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 4; 2 Hours Post-dose: number analyzed (Participants) | 1
  Cycle 4; 2 Hours Post-dose | 1290 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 4; 4 Hours Post-dose: number analyzed (Participants) | 8
  Cycle 4; 4 Hours Post-dose | 1040 (668)
  Cycle 4; 8 Hours, Post-dose: number analyzed (Participants) | 1
  Cycle 4; 8 Hours, Post-dose | 978 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 4; 24 Hours Post-dose: number analyzed (Participants) | 1
  Cycle 4; 24 Hours Post-dose | 660 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 4; 96 Hours: number analyzed (Participants) | 1
  Cycle 4; 96 Hours | 773 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 4; 168 Hours: number analyzed (Participants) | 1
  Cycle 4; 168 Hours | 767 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 4; 336 Hours: number analyzed (Participants) | 1
  Cycle 4; 336 Hours | 924 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 8; Pre-dose: number analyzed (Participants) | 4
  Cycle 8; Pre-dose | 342 (123)
  Cycle 8; 4 Hours post-dose: number analyzed (Participants) | 4
  Cycle 8; 4 Hours post-dose | 602 (290)

27. Secondary Outcome: Stage 1: Cohort 3: Plasma Concentration of Niraparib Following Niraparib Monotherapy
Description: Blood samples were collected at indicated time points.
Time Frame: Cycle 1 Day 1 (Pre-dose and 4 Hours Post-dose), Cycles 2, 4 and 8 (Pre-dose and 4 Hours Post-dose) (each cycle of 21 days)
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Stage 1 (Cohort 3): Niraparib
Number analyzed (Participants) | 3
Nanograms per milliliter
  Cycle 1 Day 1; Pre-dose: number analyzed (Participants) | 1
  Cycle 1 Day 1; Pre-dose | NA (NA) — NA indicates that data was not available as no concentration values detected for pre-dose.
  Cycle 1 Day 1; 4 Hours Post-dose: number analyzed (Participants) | 1
  Cycle 1 Day 1; 4 Hours Post-dose | 279 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 2; Pre-dose: number analyzed (Participants) | 2
  Cycle 2; Pre-dose | 469 (NA) — NA indicates that standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.
  Cycle 2; 4 Hours Post-dose: number analyzed (Participants) | 2
  Cycle 2; 4 Hours Post-dose | 717 (NA) — NA indicates that standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.
  Cycle 4; Pre-dose: number analyzed (Participants) | 1
  Cycle 4; Pre-dose | 615 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 4; 4 Hours Post-dose: number analyzed (Participants) | 1
  Cycle 4; 4 Hours Post-dose | 871 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 8; Pre-dose: number analyzed (Participants) | 1
  Cycle 8; Pre-dose | 478 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Cycle 8; 4 Hours Post-dose: number analyzed (Participants) | 1
  Cycle 8; 4 Hours Post-dose | 913 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.

28. Secondary Outcome: Stage 2: Cohorts 1A and 2A: Plasma Concentration of Niraparib Following Combination Therapy of Niraparib and TSR-042 (Dostarlimab)
Description: Blood samples were collected at indicated time points.
Time Frame: Cycle 1 Day 1 (Pre-dose and 4 Hours Post-dose), Cycles 2, 4 and 9 (Pre-dose and 4 Hours Post-dose) (each cycle of 21 days)
Population: Pharmacokinetic Population. Data was not collected for Cohort 2A of Stage 2 as no participant was enrolled into this Cohort of the study. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Stage 2 (Cohort 1A): Niraparib + TSR-042 (Dostarlimab) | Stage 2 (Cohort 2A): Niraparib + TSR-042 (Dostarlimab)
Number analyzed (Participants) | 12 | 0
Nanograms per milliliter
  Cycle 1 Day 1; Pre-dose | NA (NA) — NA indicates that data was not available as no concentration values detected for pre-dose. |
  Cycle 1 Day 1; 4 Hours Post-dose | 328 (254) |
  Cycle 2; Pre-dose: number analyzed (Participants) | 9 | 0
  Cycle 2; Pre-dose | 669 (503) |
  Cycle 2; 4 Hours Post-dose: number analyzed (Participants) | 9 | 0
  Cycle 2; 4 Hours Post-dose | 967 (540) |
  Cycle 4; Pre-dose: number analyzed (Participants) | 8 | 0
  Cycle 4; Pre-dose | 486 (243) |
  Cycle 4; 4 Hours Post-dose: number analyzed (Participants) | 8 | 0
  Cycle 4; 4 Hours Post-dose | 795 (228) |
  Cycle 9; Pre-dose: number analyzed (Participants) | 5 | 0
  Cycle 9; Pre-dose | 456 (134) |
  Cycle 9; 4 Hours Post-dose: number analyzed (Participants) | 4 | 0
  Cycle 9; 4 Hours Post-dose | 766 (231) |

29. Other Pre Specified Outcome: Stage 1: Cohort 1: Overall Survival (OS)
Description: Overall survival was defined as the time from date of first dose to the date of death due to any cause.
Time Frame: Up to a maximum of 45 months
Population: mITT Population. OS was removed as a secondary endpoint through a protocol amendment, following completion of the primary endpoint. OS will not be analyzed and reported for this study.
Arm/Group | Stage 1 (Cohort 1): Niraparib + Pembrolizumab
Number analyzed (Participants) | 0

30. Other Pre Specified Outcome: Stage 1: Cohort 2: Overall Survival
Description: Overall survival was defined as the time from date of first dose to the date of death due to any cause.
Time Frame: Up to a maximum of 17 months
Population: as for outcome 29
Arm/Group | Stage 1 (Cohort 2): Niraparib + Pembrolizumab
Number analyzed (Participants) | 0

31. Other Pre Specified Outcome: Stage 1: Cohort 3: Overall Survival
Description: Overall survival was defined as the time from date of first dose to the date of death due to any cause.
Time Frame: Up to a maximum of 6 months
Population: as for outcome 29
Arm/Group | Stage 1 (Cohort 3): Niraparib
Number analyzed (Participants) | 0

32. Other Pre Specified Outcome: Stage 2: Cohorts 1A and 2A: Overall Survival
Description: Overall survival was defined as the time from date of first dose to the date of death due to any cause.
Time Frame: Up to a maximum of 29 months
Population: as for outcome 29
Arm/Group | Stage 2 (Cohort 1A): Niraparib + TSR-042 (Dostarlimab) | Stage 2 (Cohort 2A): Niraparib + TSR-042 (Dostarlimab)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality serious adverse events (SAE) and non-SAE were collected up to a maximum of 45 months in Cohort 1-Stage 1,up to a maximum of 17 months in Cohort 2-Stage 1,up to a maximum of 6 months in Cohort 3-Stage 1 and up to a maximum of 29 months in Cohort 1A-Stage 2.
Description: Safety Population comprised of participants who received at least one dose of either study medication. Data was not collected for Cohort 2A-Stage 2 as no participant was enrolled in this Cohort.
Arm/Group | Stage 1 (Cohort 1): Niraparib + Pembrolizumab | Stage 1 (Cohort 2): Niraparib + Pembrolizumab | Stage 1 (Cohort 3): Niraparib | Stage 2 (Cohort 1A): Niraparib + TSR-042 (Dostarlimab) | Stage 2 (Cohort 2A): Niraparib + TSR-042 (Dostarlimab)
All-Cause Mortality (participants affected / at risk) | 11/17 | 16/21 | 1/3 | 6/12 | 0/0
Serious Adverse Events (participants affected / at risk) | 11/17 | 14/21 | 1/3 | 7/12 | 0/0
Other Adverse Events (participants affected / at risk) | 17/17 | 20/21 | 3/3 | 12/12 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 (Cohort 1): Niraparib + Pembrolizumab (N=17) | Stage 1 (Cohort 2): Niraparib + Pembrolizumab (N=21) | Stage 1 (Cohort 3): Niraparib (N=3) | Stage 2 (Cohort 1A): Niraparib + TSR-042 (Dostarlimab) (N=12) | Stage 2 (Cohort 2A): Niraparib + TSR-042 (Dostarlimab) (N=0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 0
Pneumonia (Infections and infestations) | 3 | 3 | 0 | 2 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 (Cohort 1): Niraparib + Pembrolizumab (N=17) | Stage 1 (Cohort 2): Niraparib + Pembrolizumab (N=21) | Stage 1 (Cohort 3): Niraparib (N=3) | Stage 2 (Cohort 1A): Niraparib + TSR-042 (Dostarlimab) (N=12) | Stage 2 (Cohort 2A): Niraparib + TSR-042 (Dostarlimab) (N=0)
Nausea (Gastrointestinal disorders) | 7 | 12 | 2 | 7 | 0
Constipation (Gastrointestinal disorders) | 7 | 10 | 1 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 0 | 6 | 0
Vomiting (Gastrointestinal disorders) | 3 | 5 | 1 | 3 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 5 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 1 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0
Fatigue (General disorders) | 8 | 9 | 1 | 5 | 0
Oedema peripheral (General disorders) | 2 | 5 | 0 | 5 | 0
Chills (General disorders) | 1 | 3 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 2 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 2 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 2 | 0 | 1 | 0
Pain (General disorders) | 0 | 3 | 1 | 1 | 0
Pyrexia (General disorders) | 2 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 0 | 2 | 0
Candida infection (Infections and infestations) | 2 | 1 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 11 | 1 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 2 | 5 | 0 | 2 | 0
Weight decreased (Investigations) | 2 | 3 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 4 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 2 | 1 | 3 | 0
Neutrophil count decreased (Investigations) | 1 | 3 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2 | 0 | 0 | 0
Amylase increased (Investigations) | 2 | 1 | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 2 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 10 | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 4 | 1 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 3 | 0 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 4 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 4 | 2 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 0 | 0 | 1 | NA
Depression (Psychiatric disorders) | 1 | 2 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 4 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 1 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 3 | 0
Hypothyroidism (Endocrine disorders) | 0 | 2 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Catheter site irritation (General disorders) | 0 | 0 | 0 | 1 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 1 | 0
Physical deconditioning (General disorders) | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Levator syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Lip disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Vitamin D decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Horner's syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatobiliary disease (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Calculus prostatic (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Penile pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Prostatic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Immobile (Social circumstances) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT03308942/Prot_002.pdf
  • Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT03308942/SAP_003.pdf